CLINICAL TRIAL: NCT00188578
Title: A Pilot Study of Conformal Intensity Modulated Radiation Therapy (IMRT) for Gynaecological Cancer Patients Not Suitable for Intracavitary Brachytherapy Boost (GY03.2)
Brief Title: Intensity Modulated Radiation Therapy - Gyne Cancer (GY03.2)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 03-0298-C
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Cervix Neoplasms; Uterine Neoplasms; Vaginal Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms; Vaginal Neoplasms

ARMS (1):
- IMRT Gynecological Cancers (Experimental)
  Interventions: Procedure: Intensity Modulated Radiation Therapy Boost

INTERVENTIONS:
Procedure: Intensity Modulated Radiation Therapy Boost — All patients shall receive a continuous course of IMRT consisting of 25.2 Gy in 14 fractions over 3 weeks

SUMMARY:
Standard treatment for gynecological cancer is radiation therapy in two phases; whole pelvic radiation and then an internal radiation boost, also called a brachytherapy boost, to treat any remaining tumour.

The purpose of this study is to test an alternative radiation boost treatment called conformal intensity modulated radiation therapy or IMRT. Currently, we do not have complete information on the overall effectiveness of IMRT compared to brachytherapy or conformal radiotherapy. We know that IMRT allows the radiation beams to be more accurately focused on the tumor, thereby sparing more normal tissue from radiation damage and lowering risks of side effects. We are investigating the extent to which IMRT can be used to protect normal tissues in patients with cervix, uterine or vaginal cancer from the radiation beams and how much the side effects of radiation are reduced.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven carcinoma of the cervix, uterus or vagina; FIGO stage T1B-4A, NO/1, MO, treated with definitive radiotherapy with or without chemotherapy, or Biopsy-proven pelvic recurrence of carcinoma of the uterus previously untreated or biopsy-proven vaginal carcinoma treated radically with radiotherapy but unsuitable for brachytherapy boost.
* Patients not suitable for intracavitary brachytherapy.
* ECOG performance status of 0, 1, or 2
* Age ≥ 18 years
* Ability to give informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of using IMRT to boost the primary tumour in patients with gynecological cancers who are unsuitable for brachytherapy. | 5 years

SECONDARY OUTCOMES:
To evaluate the acute and late toxicity of IMRT boost. | 5 years
To evaluate tumour response and patient survival data. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Fyles, MD, Principal Investigator — Princess Margaret Hospital, Canada; Michael Milosevic, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada